CLINICAL TRIAL: NCT05236439
Title: Monocentre, Non-Randomised Clinical Study Evaluating the Efficacy and Safety of Supraflow v2.2 in Glaucoma Surgery
Brief Title: Study of a Cilioscleral Interposition Device (CID) SV22 in Patients With Primary Open Angle Glaucoma and Narrow Angle Glaucoma
Acronym: SAFARI 3
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ciliatech (Industry)
Collaborators: Clinchoice Inc (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAFARI 3
Record Dates: First submitted 2022-02-02; First posted 2022-02-11 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Glaucoma, Open-Angle; Glaucoma, Narrow Angle
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma, Angle-Closure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interposition supraciliary implant (Experimental): Any patients corresponding to inclusion / exclusion criteria
  Interventions: Device: Interposition supraciliary implant

INTERVENTIONS:
Device: Interposition supraciliary implant — Surgical placement of SV22 interposition supraciliary implant in the supraciliary space

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of implanting a new version of an interposition supraciliary implant (SV22) as a stand-alone therapy for lowering intraocular pressure (IOP) in patients with primary open angle glaucoma (POAG) and primary narrow angle glaucoma (PNAG) who have failed at least one class of topical medical therapy

DETAILED DESCRIPTION:
57 patients will be included in this 36 months interventional study.

All patients shall be indicated for glaucoma surgery alone (not combined with cataract), and will undergo incisional glaucoma therapy, including a simplified surgical technique allowing the placement of an interposition supraciliary permanent device.

Several patient data like safety events, IOP, visual capacity or associated pharmacological treatments will be recorded pre and post-operatively all along the follow-up.

Purpose is to ensure device safety, and verify IOP and associated pharmacological treatment reduction after surgery, and evolution along follow-up.

ELIGIBILITY:
Inclusion criteria

To be included in the study, all patients must meet all the following inclusion criteria:

Patient:

1. 18 years or older
2. Able to understand study requirements
3. Able and willing:

   To provide written consent on the EC-approved Informed Consent Form, b. To comply with all study requirements, including required study follow-up visits' agenda

   Eye:
4. Primary Open Angle Glaucoma (POAG) or Narrow Angle Glaucoma (PNAG), including pseudo exfoliative and pigmentary glaucoma, which meets the following:

   1. Vertical C/D ratio on fundoscopic exam ≤ 0.9, or OCT demonstrating a thinness of the nerve fibre layer at the p<5% level as defined by the instrument's built in age-adjusted normative database,
   2. Glaucoma visual field (Humphrey) with -15 < MD < 0dB
5. Pharmacological treatments: glaucoma not adequately controlled by 1 to 4 different IOP-lowering medication(s), given each for at least one month prior to Screening,
6. IOP: if using 1 to 4 IOP-lowering medication, IOP is between 21 mmHg and 35 mmHg in the study eye at Screening and Baseline visits
7. Having the indication for glaucoma surgery alone (no concomitant cataract surgery)
8. Central Corneal Thickness between 480 to 620 µm
9. Gonioscopy confirming normal angle anatomy at site of implantation

Exclusion criteria

Patients will not participate in this clinical study if they meet any of the following criteria:

Patient:

1. Patient with a known allergy to any of the constituents of the products used in this study or known steroid responder
2. Patient already included in another study
3. A person protected by law (temporary or permanent guardianship) or not capable of discernment
4. Patient who may not assist to all follow-up visits (because of frequent travelling, or living in remote area, or limited moving capacities, …)
5. Pregnant or nursing woman at the date of inclusion (only for women of childbearing potential: positive urine pregnancy test at screening)
6. With uncontrolled systemic disease that, in the opinion of the Investigator, would put the subject's health at risk and/or prevent the subject from completing all study visits (e.g. inability to reliably complete visual field testing over the course of the study, or take glaucoma medications (e.g. Parkinson's disease), or uncontrolled systemic disease (diabetes, hypertension) that could compromise participation in the study, …)
7. Who have a new or modified prescription for a systemic treatment that could influence IOP within one month prior to inclusion, or who are aware of a future change in their systemic treatment, or if their medical condition indicates that their systemic treatment may change in the future
8. Chemotherapy in the last 6 months before surgery

   Eye:
9. Inflammatory, congenital, malignant, traumatic, uveitic, neovascular glaucoma or iridocorneal endothelial syndrome (ICE syndrome)
10. History of any incisional glaucoma surgery or implantable glaucoma device
11. Prior SLT, ALT or MLT
12. Eye surgery (other than glaucoma) less than 6 months ago, or presenting sequelae of previous eye surgery or trauma
13. Inability to obtain accurate IOP measurement throughout the study (e.g. history of corneal surgery, corneal opacities or disease/pathology)
14. Conditions associated with elevated episcleral venous pressure such as active thyroid orbitopathy, cavernous sinus fistula, Sturge-Weber syndrome, orbital tumors, orbital congestive disease
15. Any known ocular condition that may require intraocular intervention during the protocol required follow-up period
16. Premature or mature cataract (initial cataract are accepted)
17. Any condition that prevents the investigational device implantation in the superior and nasal region of the eye
18. Pre-existing ocular or systemic pathology that may, in the opinion of the Investigator, cause post-operative complications
19. Non laser retinal surgery
20. Previous cyclodestructive or scleral buckling procedure
21. History of complicated cataract surgery (as posterior capsular rupture, vitreous loss)
22. History of silicone oil
23. Ocular steroid in the planned study eye or systemic steroid use in the last 3 months before surgery
24. Use of oral hypotensive glaucoma medications for treatment of the fellow eye
25. Axial length <20 mm
26. Severe myopia
27. Best corrected distant visual acuity of 0.1 (20/200) or worse in the study or fellow eye
28. Peripheral synechia at the angle
29. Closed angle
30. Peripheral laser iridotomy in the last 7 days before planned surgery
31. Epithelial or fibrous downgrowth
32. Severe dry eye syndrome
33. Severe blepharitis
34. Chronic or recurrent uveitis
35. Conjunctiva showing keratitis, fine conjunctiva, erosion or abnormal vascularisation
36. Active iris neovascularization, rubeosis, proliferative retinopathy, diagnosed degenerative visual disorders (e.g. macular degeneration or other retinal disorders), vitreous haemorrhage, preretinal haemorrhage, choroidopathy or other ophthalmic disease that could confound study results
37. Scleral fixation IOL
38. Lens dislocation or subluxation
39. Vitreous loss in the anterior chamber

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2025-02-19 (Actual); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Assess post-op IOP and IOP lowering pharmacological treatments | 24 months
  Mean change in medicated IOP and IOP-lowering pharmacological treatments from baseline at 24 months after surgery

SECONDARY OUTCOMES:
Assess post op mean diurnal IOP | up to 36 months
  Proportion of eyes with ≥ 20% decrease in mean-Diurnal-IOP from baseline up to 6, 12, 18, 24 and 36 months post-operatively with IOP lowering medication
Assess mean medicated IOP | Up to 36 months
  Mean medicated IOP at Baseline and 6, 12, 18, 24 and 36 months after surgery
Mean number of IOP lowering pharmacological treatments | Up to 36 months
  Mean number of IOP-lowering pharmacological treatments at baseline and 6, 12, 18, 24 and 36 months after surgery
Mean change in post op IOP and IOP lowering pharmacological treatment | 6, 12, 18, and 36 months
  Mean change in medicated IOP and IOP-lowering pharmacological treatments from baseline at 6, 12, 18 and 36 months after surgery
Assess absolute success rate | Up to 36 months
  Absolute success rate: proportion of med-free eyes with ≥ 20% decrease from baseline and below 18 mmHg at 6, 12, 18, 24 and 36 months after surgery
Assess qualified success rate | Up to 36 months
  Qualified success rate: proportion of eyes with ≥ 20% decrease from baseline and below 18 mmHg at 6, 12, 18, 24 and 36 months after surgery
Rate of patients with a reduction in post operative IOP | Up to 36 months
  Rate of patients with at least a 20%, 30%, 40% and more than 50% reduction in post operative IOP, with or without combined medical treatments, at each visit
Proportion of eyes free of ocular hypotensive medications | Up to 36 months
  Proportion of eyes free of ocular hypotensive medications at 6, 12, 18, 24 and 36 months after surgery
Assess proportion of eyes with IOP between 6-18 mmHg | Up to 36 months
  Proportion of eyes with IOP ≥6 mmHg and ≤ 18 mmHg, the same with med-free eyes only
Proportion of eyes with IOP between 6-16 mmHg | Up to 36 months
  Proportion of eyes with IOP ≥6 mmHg and ≤ 16 mmHg, the same with med-free eyes only
Average number of adjunctive therapies post-operatively | Up to 36 months
  Average number of adjunctive therapies (needling, goniopuncture, SLT, …) performed up to 36 months postoperatively
Rate of patients with no filtering blebs | Up to 36 months
  Rate of patients with no filtering bleb, average duration of filtering blebs
Assess the surgical procedure | Day 0, day of surgery
  To evaluate the surgical procedure (duration of operation, ease of implantation)
Assess patient satisfaction post-operatively | Up to 36 months
  To describe patient satisfaction following surgery based on criteria of pain, discomfort and deterioration in visual acuity
Describe patient's quality of life | Up to 36 months
  To describe changes in quality of life (EQ5D)
Assess rate of intraoperative and post-operative related adverse device effects | Up to 36 months
  Rate of intraoperative and post-operative device related ocular adverse events and adverse device effect
Review slit lamp, gonioscopy and fundus findings | Up to 36 months
  Slit lamp, gonioscopy and fundus findings
Determine rate of BCVA | Up to 36 months
  Rate of best corrected visual acuity variation (BCVA)
Assess rate of Visual field mean deviation variation (VF MD) | Up to 36 months
  Rate of Visual field mean deviation variation (VF MD)
Determine rate of C/D ratio mean deviation | Up to 36 months
  Rate of C/D ratio mean deviation
Assess rate of sight threatening events | Up to 36 months
  Rate of sight threatening events
Assess rate of change in endothelial cell density and central corneal thickness | Up to 36 months
  Rate of change in endothelial cell density (ECD) and central corneal thickness (CCT)
Assess rate of occurrence of SV22 movements in the supraciliary space | Up to 36 months
  Rate of occurrence of SV22 movements inside the supraciliary space (SCS), defined as a change of position of the anterior edge of the implant of at least 200 µm measured on UBM from D7 to any timepoint

CONTACTS AND LOCATIONS:
Overall Officials: Lilit Voskanyan, Principal Investigator — Malayan Center
Locations (1):
- Malayan center, Yerevan, Yerevan, Armenia

IPD SHARING:
Plan to Share IPD: No